CLINICAL TRIAL: NCT07398144
Title: Laparoscopic Burch Colposuspension Versus Transobturator Tape in the Treatment of Female Stress Urinary Incontinence. A Prospective Randomized Study
Brief Title: Laparoscopic Burch Colposuspension Versus Transobturator Tape in the Treatment of Female Stress Urinary Incontinence.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Theodor Bilharz Research Institute (Other)
Responsible Party: Principal Investigator, Mohamed Fathi Mohamed Ahmed Badr-El-Din, Urology specialist, Theodor Bilharz Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MD-94-2025
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Female Stress Urinary Incontinence
Keywords: laparoscopic Burch; trans obturator tape; TOT; Female Stress Urinary Incontinence; colposuspension; SUI; stress urinary incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A laparoscopic Burch (Active Comparator): laparoscopic Burch colposuspension
  Interventions: Procedure: laparoscopic Burch colposuspension
- group B TOT (Active Comparator): Trans obturator tape
  Interventions: Procedure: Trans obturator tape fixation

INTERVENTIONS:
Procedure: laparoscopic Burch colposuspension — laparoscopic Burch colposuspension for female stress urinary incontinence
  Arms: group A laparoscopic Burch
Procedure: Trans obturator tape fixation — mid urethral sling for female stress urinary incontinence
  Arms: group B TOT

SUMMARY:
The goal of this prospective interventional study is to compare the effectiveness of laparoscopic Burch colposuspension versus trans obturator tape in the treatment of stress urinary incontinence in adult females. The success rate will be compared between the two proceudres at 1, 3 and 6 months post operatively. Operative times, hospital stay and perioperative complications will be evaluated in both arms

Participants will be asked to:

* complete the ICIQ-UI-SF questionnaire pre operatively and at 1, 3 and 6 months post operatively
* undergo a pelvic examination pre operatively
* undergo cough stress test pre operatively and at 1, 3 and 6 months post operatively
* undergo a pressure flow study test pre operatively
* undergo pelviabdominal ultrasound with post void residual urine measurement pre operatively and at 1, 3 and 6 months post operatively
* undergo uroflowmetry at 1 month post operatively

DETAILED DESCRIPTION:
This is a prospective randomized study that is conducted at Theodor Bilharz research institute and Cairo university hospital. the study will include 60 female patients with genuine stress urinary incontinence allocated randomly to 2 groups; group A will undergo laparoscopic Burch colposuspension and group B which will undergo trans obturator tape fixation.

The investigators aim to evaluate the success rates of laparoscopic Burch colposuspension and TOT procedures in treatment of female SUI. Objective cure rates, assessed by cough stress test or pad weight test. ( A cure is defined as the absence of a subjective complaint of leakage and the absence of objective leakage during a 250-ml cough stress test. operation time and length of hospital stay as well as early outcomes, complications and continence rates at 1 month, 3 months and 6 months will be recorded and compared.

Inclusion criteria:

• Clinical Diagnosis of SUI: Symptoms include leakage during activities such as coughing, sneezing, laughing, or physical exertion.

* Documented stress urinary incontinence by physical examination and urodynamic testing.
* Adult female patients typically aged 18 years or older.
* Completed Non-Surgical Management:

Patients who have tried and failed conservative management options, such as pelvic floor exercises, behavioral therapy.

• Willingness to Undergo Surgery

Exclusion criteria:

* Mixed urinary Incontinence
* Pelvic Organ Prolapse more than the 2nd degree according to Baden and Walker classification 1992
* Previous Anti-Incontinence Surgery
* Neurological Conditions:

Patients with neurogenic bladder or other neurologic disorders affecting bladder function, such as multiple sclerosis or spinal cord injury.

* Pregnancy
* Presence of active urinary tract infection (UTI) or other pelvic infections at the time of evaluation
* Patients with interstitial cystitis, bladder tumors, or urethral diverticula that could complicate surgical outcomes
* Previous history of radiotherapy to the pelvis.
* Contraindications to surgery such as uncorrectable coagulation disorders

Methodology All patients will provide oral and written consent before participating in any study-related procedures.

Preoperative Assessment:

* History ((using validated questionnaire (International Consultation on Incontinence Questionnaire- Urinary Incontinence Short Form (ICIQ-UI SF) and physical examination to confirm stress incontinence and exclude overactive bladder syndrome.
* Pelvic examination to rule out pelvic organ prolapse.
* Routine preoperative labs (CBC, coagulation profile, electrolytes)
* Urodynamic studies to confirm SUI
* Pelvi-abdominal Ultrasonography to measure PVR.
* Urine culture and sensitivity to exclude urinary tract infection. post operative work up:
* Catheter removal after 24 hours.and monitoring for urine retention and catheterization if required
* follow up scheduled at 1 month, 3 months and 6 months postoperatively targeting success rate, PVR and complications. (uroflowmetry at 1 month-visit)

Primary Outcomes:

Objective cure rates, assessed by cough stress test or pad weight test ( we use the pad test when the cough test is negative but the patient reports leakage during daily activities or patient is still has leakage after operation to compare the number of pads preoperatively and post-operatively ). ( A cure is defined as the absence of a subjective complaint of leakage and the absence of objective leakage during a 250-ml cough stress test.)

Secondary Outcomes:

* Improvement in SUI symptoms (e.g., using validated questionnaires (International Consultation on Incontinence Questionnaire).
* Comparing Peri-operative and early outcomes (e.g. hemoglobin loss, operation time, and length of hospital stay.).
* Intraoperative and early complications (e.g. Bladder injury, infection, De novo urge incontinence, and Acute Urinary Retention, post-void residual volume).

ELIGIBILITY:
Inclusion Criteria:

* Clinical Diagnosis of SUI:

Symptoms include leakage during activities such as coughing, sneezing, laughing, or physical exertion.

* Documented stress urinary incontinence by physical examination and urodynamic testing.
* Adult female patients typically aged 18 years or older.
* Completed Non-Surgical Management:

Patients who have tried and failed conservative management options, such as pelvic floor exercises, behavioral therapy.

• Willingness to Undergo Surgery

Exclusion Criteria:

* virgin female
* mixed urinary Incontinence

  * Pelvic Organ Prolapse more than the 2nd degree according to Baden and Walker classification 1992
  * Previous Anti-Incontinence Surgery
  * Neurological Conditions:

Patients with neurogenic bladder or other neurologic disorders affecting bladder function, such as multiple sclerosis or spinal cord injury.

* Pregnancy
* Presence of active urinary tract infection (UTI) or other pelvic infections at the time of evaluation
* Patients with interstitial cystitis, bladder tumors, or urethral diverticula that could complicate surgical outcomes
* Previous history of radiotherapy to the pelvis.
* Contraindications to surgery such as uncorrectable coagulation disorders

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-01-02 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
success rate | at 1, 3 and 6 months post operative
  the absence of a subjective complaint of leakage and the absence of objective leakage during a 250-ml cough stress test

SECONDARY OUTCOMES:
operative time | day 1 post operative
complicatio rate | till 6 months post operative
hospital stay | 2 days post operative

CONTACTS AND LOCATIONS:
Overall Officials: Hussein A Hussein, professor of urology, Study Director — professor of urology , Faculty of medicine , Cairo university; Ahmed I Kamel, professor of urology, Study Chair — professor of urology , Theodor Bilharz Research Institute; Ahmed H Abo-Zamel, assistant professor of urology, Study Chair — assistant professor of urology , Faculty of medicine , Cairo university; Ahmed S Kamel, lecturer of urology, Study Chair — lecturer of urology , Faculty of medicine , Cairo university
Locations (2):
- Egypt (2):
  - Cairo university hospitals, Giza, Giza Governorate
  - Theodor Bilharz Research Institute, Giza, Giza Governorate

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: all the IPD will be available from date of publication and for 6 months
Access Criteria: All urologists and gynecologists interested in stress incontinence via the contact information of the principle investigator

REFERENCES:
- [Result] Freites J, Stewart F, Omar MI, Mashayekhi A, Agur WI. Laparoscopic colposuspension for urinary incontinence in women. Cochrane Database Syst Rev. 2019 Dec 10;12(12):CD002239. doi: 10.1002/14651858.CD002239.pub4. PMID 31821550
- [Result] Brasoveanu S, Balulescu L, Grigoras D, Erdelean D, Olaru F, Bardan R, Balint O, Margan MM, Alexandru A, Cristiana-Smaranda I, Pirtea L. Evaluating Patient Preferences and Clinical Outcomes for Modified Laparoscopic Burch Colposuspension and Transobturator Tape Procedures in Stress Urinary Incontinence Treatment. Life (Basel). 2024 Mar 14;14(3):380. doi: 10.3390/life14030380. PMID 38541705
- [Result] D'Ancona C, Haylen B, Oelke M, Abranches-Monteiro L, Arnold E, Goldman H, Hamid R, Homma Y, Marcelissen T, Rademakers K, Schizas A, Singla A, Soto I, Tse V, de Wachter S, Herschorn S; Standardisation Steering Committee ICS and the ICS Working Group on Terminology for Male Lower Urinary Tract & Pelvic Floor Symptoms and Dysfunction. The International Continence Society (ICS) report on the terminology for adult male lower urinary tract and pelvic floor symptoms and dysfunction. Neurourol Urodyn. 2019 Feb;38(2):433-477. doi: 10.1002/nau.23897. Epub 2019 Jan 25. PMID 30681183